CLINICAL TRIAL: NCT00267553
Title: Open Label Treatment and Survival Continuation Study of Atamestane Plus Toremifene Versus Letrozole in Advanced Breast Cancer
Brief Title: Treatment and Survival Continuation Study of Atamestane Plus Toremifene vs Letrozole in Advanced Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This was a follow-on study to Biomed 777-CLP-029 which did not meet superiority endpoint
Sponsor: Intarcia Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Biomed 777-CLP-32
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Breast Neoplasms; Neoplasms, Hormone-Dependent
Keywords: Atamestane; Breast neoplasms; Combined hormonal therapy; Complete estrogen blockade; Ductal breast carcinoma; Estrogen blocker; Fareston®; Femara®; First line therapy; Letrozole; Lobular breast carcinoma; Locally advanced breast cancer; Locally recurrent breast cancer; Maximal estrogen inhibition; Metastatic breast cancer; Neoplasms, Hormone-dependent; Receptor-positive; Stage IIIA breast cancer; Stage IIIB breast cancer; Stage IV breast cancer; Toremifene
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Hormone-Dependent; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — atamestane; Toremifene; Letrozole

INTERVENTIONS:
Drug: Atamestane
Drug: toremifene
Drug: letrozole

SUMMARY:
Protocol 777-CLP-32 is the treatment and survival continuation protocol of Biomed 777-CLP-29, and will continue to compare combined hormonal therapy using the experimental aromatase inhibitor (AI) atamestane combined with the FDA-approved anti-estrogen toremifene (Fareston®), to the single agent FDA-approved aromatase inhibitor letrozole (Femara®) for the treatment of advanced breast cancer. The purpose of this study is to determine whether maximal estrogen suppression achieved via the combination of atamestane, plus toremifene (Fareston®), is more effective than letrozole (Femara®) in delaying the growth of breast cancer.

DETAILED DESCRIPTION:
Aromatase is an enzyme expressed in tissues such as muscle and fat in postmenopausal women. These non-ovarian tissues become the dominant sources of estrogen in postmenopausal women. Breast cancer cells are often very dependent on estrogens to continue to grow. Atamestane blocks the formation of estrogens from androgenic precursors in the body via the aromatase enzyme. Toremifene blocks circulating and intracellular estrogens from stimulating estrogen receptors in breast cancer cells. The goal of therapy with atamestane, an aromatase inhibitor, in combination with the estrogen receptor antagonist, toremifene, is to achieve complete suppression of estrogen stimulation of breast cancer cells. This study is designed to determine whether combined hormonal therapy will lengthen the time to disease progression and the survival time for subjects with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to receive continued treatment, subjects must remain eligible to receive study drug at the time of their last Biomed 777-CLP-29 visit
* To continue on survival follow-up, subjects must be in survival follow-up in study Biomed 777-CLP-29
* Written informed consent obtained for subjects who continue study drug treatment

Exclusion Criteria:

* Subjects who have withdrawn consent to participate in Biomed 777-CLP-29 for any reason
* Subjects for whom the investigator considers study participation is no longer in the best interest of those subjects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
In conjunction with the data from Biomed 777-CLP-29, compare the time to progression (TTP) in the atamestane plus toremifene arm to the TTP in the letrozole plus placebo arm

SECONDARY OUTCOMES:
In conjunction with the data from Biomed 777-CLP-29, obtain safety, survival and time to treatment failure (TTF) data for both arms in this continuation study.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langecker, MD, PhD, Study Director — Intarcia Therapeutics
Locations (35):
- United States (6):
  - Greenbrae, California
  - Saint Joseph, Michigan
  - Kansas City, Missouri
  - Houston, Texas
  - Norfolk, Virginia
  - Lacey, Washington
- Canada (3):
  - Ottawa, Ontario
  - Thunder Bay, Ontario
  - Montreal, Quebec
- Russia (17):
  - Arkhangelsk
  - Kazan'
  - Krasnodar
  - Leningrad Region
  - Lipetsk
  - Moscow
  - Murmansk
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Stavropol
  - Tomsk
  - Veliky Novgorod
  - Voronezh
- Ukraine (9):
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kryvyi Rih
  - Lviv
  - Odesa
  - Uzhhorod